CLINICAL TRIAL: NCT00312143
Title: A Prospective, Open Label, Multicenter Study to Assess the Efficacy and Safety of Enteric-coated Mycophenolate Sodium (EC-MPS) in de Novo Kidney Transplant Recipients
Brief Title: Efficacy and Safety of Enteric-coated Mycophenolate Sodium (EC-MPS) in de Novo Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CERL080AEG01
Record Dates: First submitted 2006-04-05; First posted 2006-04-07 (Estimated); Last update posted 2011-02-02 (Estimated); Status verified 2011-02

CONDITIONS: De Novo Kidney Transplant Recipients
Keywords: De novo Kidney Transplant recipients, enteric-coated mycophenolate sodium

INTERVENTIONS:
Drug: Enteric-coated Mycophenolate sodium (EC-MPS)

SUMMARY:
This trial is designed to assess the efficacy, tolerability, and safety of EC-MPS in combination with cyclosporine microemulsion (CsA-ME) with or without steroids in kidney transplant recipients.

ELIGIBILITY:
Inclusion criteria

1. Males and females aged 18 to 75 years.
2. Recipients of living related kidney transplant, treated with cyclosporine, with or without corticosteroids, as primary immunosuppression.
3. Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to or at screening. Effective contraception must be used during the trial, and for 6 weeks following discontinuation of the study medication, even where there has been a history of infertility.
4. Patients who are willing and able to participate in the full course of the study and from whom written informed consent has been obtained.

Exclusion criteria:

1. Multi-organ recipients (e.g. kidney and pancreas) or previous transplant with any organ, other than kidney.
2. Patients with any known hypersensitivity to other components of the formulation (e.g. lactose).
3. Patients with low platelet count (< 75,000/mm3), with an absolute neutrophil count of < 1,500/mm3, and/or leukocytopenia (< 2,500/mm3), and/or hemoglobin < 6 g/dL at screening or baseline.
4. Patients who have received an investigational drug within four weeks prior to study entry.
5. Patients with a history of malignancy within the last five years, except excised squamous or basal cell carcinoma of the skin.
6. Females of childbearing potential who are planning to become pregnant, who are pregnant and/or lactating, who are unwilling to use effective means of contraception.

Additional protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2004-02; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
patient and graft survival
acute rejection incidence
graft function at 6 months post transplant.

SECONDARY OUTCOMES:
influence of age, gender, and post-transplantation complications on the main clinical outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis